CLINICAL TRIAL: NCT04645186
Title: CALCIUM PHOSPHATE CEMENT AS BONE VOID FILLER - a Prospective Cohort Study in Patients Indicated for Long Bone and Extremity Surgery
Brief Title: Calcium Phosphate Cement As Bone Void Filler
Status: Terminated | Type: Observational
Why Stopped: The study was terminated following a change in company management.
Sponsor: Bioceramed (Industry)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.04
Record Dates: First submitted 2020-11-16; First posted 2020-11-27 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Bone Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Calcium Phosphate Cement (CPC): Evaluation of CPC in long bone & extremities
  Interventions: Device: bone graft substitute

INTERVENTIONS:
Device: bone graft substitute — Filling bone defects in current clinical practice

SUMMARY:
This is an observational, prospective, non-randomised, post market clinical follow-up study to compile clinical data on performance and safety of the synthetic bone graft substitute and to assess that the performance and safety of the device are maintained until the reaching of its intended use in a commercial clinical setting in long bone and extremity defects.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring bone grafting after post-traumatic or surgically created bone defects afflicting the long bones and extremities.
* Give written informed consent to participate in the study and be willing to comply with the protocol requirements.
* Able to verbalize and differentiate regarding the location and intensity of pain.
* Physical and mental availability to meet the clinical and radiographic follow-up schedule.

Exclusion Criteria:

* Serious infection within two months before surgery.
* Active malignancy, Cellulitis, Osteomyelitis, Osteomyelitis, Bone metastasis, Other bone metabolic diseases.
* Primary bone tumors and contraindications in performing an X-ray or CTscan.
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study.
* The subject is unable or not willing to complete follow-up visits and examination for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is considered as all the patients included in the study that meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Radiological healing | 3 months
  Bone healing observable by x-ray/CT-scan. Assessment of trabecular defects: modified Neer classification. Assessment of cortical defects: modified RUST.
Radiological healing | 6 months
  Bone healing observable by x-ray/CT-scan. Assessment of trabecular defects: modified Neer classification. Assessment of cortical defects: modified RUST.
Radiological healing | 9 months
  Bone healing observable by x-ray/CT-scan. Assessment of trabecular defects: modified Neer classification. Assessment of cortical defects: modified RUST.
Radiological healing | 12 months
  Bone healing observable by x-ray/CT-scan. Assessment of trabecular defects: modified Neer classification. Assessment of cortical defects: modified RUST.
Radiological healing | 18 months
  Bone healing observable by x-ray/CT-scan. Assessment of trabecular defects: modified Neer classification. Assessment of cortical defects: modified RUST.
Radiological healing | 24 months
  Bone healing observable by x-ray/CT-scan. Assessment of trabecular defects: modified Neer classification. Assessment of cortical defects: modified RUST.

SECONDARY OUTCOMES:
Number and description of any adverse event during the follow-up | 3 months
  Record and description of any adverse event during the follow-up that reflects the safety of the bone graft substitute.
Number and description of any adverse event during the follow-up | 6 months
  Record and description of any adverse event during the follow-up that reflects the safety of the bone graft substitute.
Number and description of any adverse event during the follow-up | 9 months
  Record and description of any adverse event during the follow-up that reflects the safety of the bone graft substitute.
Number and description of any adverse event during the follow-up | 12 months
  Record and description of any adverse event during the follow-up that reflects the safety of the bone graft substitute.
Number and description of any adverse event during the follow-up | 18 months
  Record and description of any adverse event during the follow-up that reflects the safety of the bone graft substitute.
Number and description of any adverse event during the follow-up | 24 months
  Record and description of any adverse event during the follow-up that reflects the safety of the bone graft substitute.

CONTACTS AND LOCATIONS:
Overall Officials: Nuno A Ribeiro, MD, Principal Investigator — Hospital Lusíadas Lisboa
Locations (1):
- Hospital Lusíadas Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No